CLINICAL TRIAL: NCT02401516
Title: Effect Of Postural Reprogramming Insoles In Regulating Blood Pressure, Posture And Quality Of Life In Hypertensive Subjects
Brief Title: Reprogramming Insoles In Regulating Blood Pressure In Hypertensive Subjects
Acronym: RIBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Bahiana de Medicina e Saude Publica (Other)
Responsible Party: Principal Investigator, ANA LUCIA BARBOSA GOES, PHYSICAL THERAPIST AND PROFESSOR AT ESCOLA BAHIANA DE MEDICINA E SAÚDE PÚBLICA, Escola Bahiana de Medicina e Saude Publica
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE 16952113.5.0000.5544
Record Dates: First submitted 2015-03-09; First posted 2015-03-30 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Hypertension
Keywords: Postural Reprogramming Insole; Blood Pressure; Posture; Quality Of Life; General Functional Capacity; Respiratory Muscles Strength; Flexibility; Arterial Systemic Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reprogramming Insoles (Active Comparator): EG - experimental group. Subjects will be subjected to the use of insoles with the artifact in the postural reprogramming insole that emits a electrogalvanic stream. Volunteers of this research must use the insole for at least 12 hours a day and have usage control through a daily chart.
  Interventions: Device: Reprogramming insoles
- Neutral Insoles (Placebo Comparator): CG - control group. Subjects will be subjected to the use of insoles likewise the ones used by EG, but instead the artifact in the postural reprogramming insole made of metal, will be made of cork.
  Interventions: Device: Reprogramming insoles

INTERVENTIONS:
Device: Reprogramming insoles — 1)Answer demographic, lifestyle and health questionnaire; 2)Weight and height evaluation; 3)ABPM (Ambulatory Blood Pressure Monitoring) and diary of activities assessment; 4)Postural Assessment software (SAPO), created by São Paulo's University (USP), which assesses posture through full body images of people with marked bone prominences on the body in all planes of motion. Images are captured by a Sony Cybershot 14 Megapixel camera, supported on a tripod, placed three meters away from the subject and at half its height. 5)Six-Minutes Walk Test in accordance with Britto and Souza25 and American Thoracic Society guidelines43; 6)analog manometer Globalmed® brand to assess respiratory muscle strength; 7)Dynamometer Jamar® brand to measure grip strength; 8)Wells bank to evaluate Flexibility.

SUMMARY:
ASH has a high prevalence rates and considered one of the major modifiable risk factors for cardiac vascular diseases (CVD) and brain vascular diseases (BVD) and one of the most important public health problems. Researches estimated 62% of BVD can be attributed to ASH. In Brazil, prevalence of hypertension ranged from 21.6% in 2006 to 42.4% in 2011. CVD are responsible for high frequency of hospitalization, and in 2009, 91,970 hospitalizations due to CVD cost public treasury more than 165 million reais. ASH neurological pathophysiology studies has shown that excessive activation of sympathetic autonomic nervous system (SANS) seems to have an important role in genesis and maintenance of ASH, with current studies aimed to understand this relationship.

Pathways used by SANS for immediate control of BP (wich are reticulate formation, bulb and cortex) appear to be similar to pathways used for postural control reflex (reticulate formation, bulb, cortex, among others), which are also used by Postural Reprogramming Insoles (PRI) for posture adequacy. Due to this similarity in reflex activation areas, it is believed that PRI may have some effect on BP regulation.

There are many ways to treat postural changes and one of them is posturology, which is based on therapeutic use of postural reprogramming insoles (PRI). PRI activates tonic-postural system, rebalancing muscles, joints and bony structures of body segments, and returning individual to an appropriate posture.

The PRI is composed of a central artifact, situated in reflex zone full of somatosensory stimuli captors, which generates a frequency of vibration that promotes postural adaptation.

DETAILED DESCRIPTION:
Posture can be defined as the way body acquires at any given time in relation to gravity line, and suffers influence of sensory information from different segments, organs and systems, integrated to cerebral cortex. Once information is associated, analyzed and compared, is sent to tonic and phasic-tonic muscles that will perform necessary adjustments to maintain posture.

When sensory information captured by body are unbalanced, body reacts to this information with deformities and misalignment like flat feet, scoliosis, among others. Posturology is a way of treating these alignment changes, which is based on use of postural reprogramming insoles (PRI) to return individual to an appropriate posture. The PRI is composed of a central artifact which stimulates autonomic system, via tonic postural system, promoting posture adaptation/regulation.

What is not known, though, is the influence of these insoles on other systems such as cardiovascular system and on other conditions, such as arterial systemic hypertension (ASH), a multifactorial clinical condition characterized by high and constant levels of blood pressure (BP).

ASH neurological pathophysiology studies has shown that excessive activation of sympathetic autonomic nervous system (SANS) seems to have an important role in genesis and maintenance of ASH, with current studies aimed to understand this relationship.

Previous studies indicate that, despite efforts to understand and control arterial systemic hypertension, rates of ASH control are low and some difficulties are listed such as: access to health services and medications, adherence to guidelines, quantity of medication usage, non-controlling hypertension even on medication, family help regarding treatment, difficulty in maintaining regular practice of physical exercise. Therefore, it is necessary to encourage dietary control, increased patient support and new forms of affordable and effective non-pharmacological treatment, in addition to measuring the impact disease causes in life and living of those patients.

Arterial Systemic Hypertension impacts physical health, psychological well-being, longevity and quality of life (QOL), and therefore should quality of life be an important criterion for studying, once it can be used as indicator of impacts that illness can provoke in individuals as well as provide data about individual adaptation.

Quality of life (QOL) is defined by WHO as the "individual's perception of their position in life in the context of culture and value systems in which they live and in relation to their goals, expectations, standards and concerns".

Health-related quality of life (HRQOL) is evaluated based on objective and measurable data, applied to sick people to identify committed dimensions and discomfort degree associated with limitation disease and/or therapy can cause. Thus, health professionals can effectively measure impact of interventions on health-related quality of life.

Instruments that assess HRQOL are usually questionnaires that must go through a validation process for language-country, in this case Portuguese.

From all HRQOL questionnaires validated in Brazil, there is one specific to assess quality of life in hypertension individuals, called Mini-Questionnaire Quality of Life in Hypertension - MINICHAL, which was developed in Spain in 2001, and validated in Brazil in 2007.

THEORETICAL RATIONALE Imbalances that affect posture are a reflection of asymmetry in Tonic Postural System (TPS). The simplified model of organization of STP states that equilibrium depends on the fascia and muscles viscoelastic system to maintain balance against body mass actions, gravity, and height.

In a standing position, fascia is not able to overcome forces opposing gravity, lonely, requiring joint muscle action to balance forces on body.

Posture can be classified as appropriate or inappropriate. When sensory information captured by body are symmetrical and well organized, tonic-postural system reaction generates minimal overload of bone, joint and myofascial structures, producing a lower energy expenditure for maintenance of these structures, favoring relative alignment to gravity and individual has an appropriated posture.

If sensory information, captured by body are unbalanced, inconsistent and disorganized, tonic-postural system requires more of muscles, joints, fascia and bone structures, to keep body segments reacting to gravity force. It creates a disharmonious relationship of various parts of body, producing a greater burden in supporting structures and a less efficient body balance on their stand weight basis, creating greater energy expenditure, misalignment and deformities like flat feet, knees valgus, scoliosis, among others and then person has poor posture.

During motion, there is a predicted movement and movement that is actually done. Between these two points there is cerebellum, which is the structure that compares predicted and performed movements by promoting postural adjustments, carried out so that movement is close to what was expected. Cerebellum organizes, provides, adjusts and modifies movement.

Adaptation system function to get body back into balance in cases of imbalance, which can be both internal and external. Terminal system adaptation is foot and therefore there is no reprogramming in TPS without focusing foot, with use of postural reprogramming insole (PRI).

PRI artifact is formed by two crossed polarizing devices, which creates a electrogalvanic field that loads and unloads, causing vibration that integrates with energy field of individual. This integration leads to a permanent posture recalibration, aligning individual in relation to gravity forces with consequent improvement of postural changes secondary to imbalances.

These sensory stimuli use SANS to stimulate areas of brain such as cerebellum, vestibular nuclei, basal nuclei (BN), reticulate formation of bulb and frontal premotor cortex to cause posture correction.

BP control is also related to SANS, which uses nerve reflex by stimulating baroreceptors, located in arteries walls and when distended, as happens in high BP, send signals to glossopharyngeal nerve and reticular formation of medulla, brain stem, causing inhibition of vasoconstrictor center and exciting vagal center, with consequent: vasodilation of veins and arterioles, decreased heart rate (HR) and heart contraction force, leading to fall reflex of BP due to decreased peripheral resistance and cardiac debit, respectively.

However, what seems to occur as shown in recent studies is the existence of a constant activation / stimulation of vasoconstrictor center in hypertensive individuals, causing BP to remain at high levels.

Stimulation of vasoconstrictor center suffers influence of SANS, which uses areas of reticulate formation, bulb and cerebral cortex, which areas appear to be similar to those used for reflex control of posture (reticulate formation, bulb, cortex, among others), which are also used by PRI for posture correction. Due to this similarity in areas of reflex activation, it is believed that PRI may have some effect on BP regulation.

Once occurring regulation of blood pressure due to use of PRI and improved posture, it is expected a positive effect on health-related quality of life of hypertensive patients.

Mini-Questionnaire Quality of Life in Hypertension - MINICHAL-Brazil suffered cultural adaptation and validation into Portuguese, which was tested for content, construct and internal consistency of instrument, comparing outcomes in hypertensive patients and patients with normal BP. Subsequently, other studies have been published testing concurrent validity by comparing Minichal with two other questionnaires used in many researches in Brazil: Short Form 36 (SF-36) and the WHOQOL questionnaire (WHOQOL-Bref), showing significant correlation to both questionnaires, making a specific tool for assessing health-related quality of life in hypertensive population.

Whereas many studies have been developed in the later stages of hypertension and impairments in functional capacity, respiratory and locomotor were observed in these stages; Whereas it is a chronic and systemic condition of progressive evolution; Whereas this study addresses a hypertensive population stage I and II without target organ injury; it is important to identify if in the early stages of this condition (stages I and II) it is possible to observe changes in above mentioned systems, identifying effects of hypertension in functional capacity, respiratory and locomotor systems, not only with character of prevention, but also for early diagnosis and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with hypertension (PAS≥140mmHg and PAD≥90mmHg), for at least two months
* Both sexes,
* Between 30-60 years;
* Living in Salvador and metropolitan area,
* Body mass index (BMI) to 29.9kg / m2,
* In regular use of anti-hypertensive drugs

Exclusion Criteria:

* Individuals with neurological diseases, mental depression, renal failure, pregnancy and diabetes mellitus associated with hypertension,
* With a history of previous cardiovascular event (myocardial infarction, heart failure, unstable angina, peripheral arterial disease)
* Undertake regular exercise

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Control by ABPM (Ambulatory Blood Pressure Monitoring) - mm Hg | Baseline and after 6 weeks insoles
  Subjects will undergo ABPM (Ambulatory Blood Pressure Monitoring), a technique that allows multiple indirect measurements of blood pressure for 24 or more consecutive hours with a minimum of discomfort during daily activities (MAPA, 2005). ABPM will be held by oscillometric method, BP measured every 15 minutes. ABPM will be used in accordance with ABPM I-II of IV Guideline tables. Subjects will also fill a diary of activities with data on symptoms and other situations that may modify BP. ABPM will be performed one day before PRI use to define baseline BP values, and six weeks after reassessment is performed using insole and is considered as endpoint the BP mean.

SECONDARY OUTCOMES:
Influence of posture alterations on blood pressure control in hypertensive individuals | Baseline
  Subjects will undergo ABPM (Ambulatory Blood Pressure Monitoring) for blood pressure measurements. Posture alterations will be observed through images taken accordingly to Postural Assessment Software (PAS) protocol.
Composite Outcome measure - Association between Blood Pressure and Posture | 6 weeks
  Verify whether there is an association between blood pressure control and improved posture.
Quality of Life domains | 6 weeks
  Identify the most common areas that impact quality of life in hypertensive subjects.
Description impact of High Blood Pressure by ABPM (Ambulatory Blood Pressure Monitoring) | Baseline and 6 weeks
  Describe General functional capacity, overall muscle strength, respiratory muscle strength and flexibility of hypertensive individuals
Compare estimated and predicted values of Six-minutes Walk Test. | Baseline
  Compare estimated and predicted values of general functional capacity in hypertensive individuals.
Compare estimated and predicted values of respiratory muscle strength. | Baseline
  Compare estimated and predicted values of breathing muscle strength in hypertensive individuals.
Changing in Posture by Postural Assessment software (SAPO) | Baseline and 6 weeks
  Postural Assessment software(SAPO), by São Paulo's University(USP), assesses posture through people full body images with marked bone prominences. Subjects wear appropriate clothing (women-shorts and tops and men-short). Hemispheres of 20-25mm diameter, colored, will be glued to bone prominences with double sided tape(3M brand) according to protocol. Feet positioned in abduction of 30° for alignment and standardization of images. After, subjects will be positioned on a plate, near a plumb line, marked 10cm length for image calibration purposes, which is attached to the ceiling. Images are captured by a Sony Cybershot 14 Megapixel camera, supported on a tripod, placed three meters away from the subject and at half its height.
  All measurements of distances are estimated in centimeters and angles in degrees.
Changing in Quality of Life by Mini-Questionnaire of Quality of Life in Hypertension: - MINICHAL-Brazil | Baseline and 6 weeks
  Questionnaire contains 16 items, 1-9 items related to Mental State dimension, with a maximum score of 27; and items 10-16 for Somatic Manifestations dimension, with a maximum score of 21 points. Questions refer to individual state in past seven days. Scoring scale is Likert-type with four possible answers: 0 = not at all; 1 = yes, a little; 2 = yes, quite; 3 = yes, very. The lower final score, the better quality of life.
Changing in General Functional Capacity using the Six-minutes Walking Test protocol | Baseline and 6 weeks
  Functional capacity of hypertensive individuals will be evaluated using the Six-minutes Walk Test which protocol will be in accordance with Britto and Souza and American Thoracic Society guidelines. Thus, subjects were instructed to walk as quickly as possible without running around a 30 meters track oriented to stop test in presence of dyspnea, severe fatigue, tachycardia and / or any other uncomfortable situation.
Changing in Overall muscle strength by dynamometer Jamar® brand to measure grip strength. | Baseline and 6 weeks
  Subjects remain seated, with both arms flexed at 90 ° and forearm in neutral rotation. Grip distance of dynamometer was individually adjusted according to hands size, so that closer shaft dynamometer body was placed on the second phalanges of the fingers: index, middle and ring finger. Resistance was graded at level II for everyone. Recovery time between measurements was about one minute. Test was performed in three attempts in hand that participant considered stronger. Best result of three attempts was used.
Changing in Respiratory muscle strength by analog manometer Globalmed® brand. | Baseline and 6 weeks
  Subjects remain seated, with elbows bent and hands firmly holding manometer nozzle near mouth. To evaluate maximum inspiratory pressure (MIP), subject will conduct maximal expiration to residual volume (RV), and after proper positioning of the equipment in the patient's mouth will be performed forced inspiration (PImax). To evaluate maximum expiratory pressure (MEP) subject will initiate from total lung capacity (TLC), followed by completion of forced expiration, noting that equipment was properly positioned in patient's mouth and adding a nose clip to prevent airflow escape. Average duration of test is about six seconds each, with one-minute interval between measurements. Will be considered for analysis the best result.
Changing in Flexibility measured through Wells bank. | Baseline and 6 weeks
  Test consists in checking trunk and posterior muscles flexibility. Subjects should sit on a hard surface, with outstretched legs and bare feet flat on the box, ankle in neutral position, one hand over other, keeping fingers together, overlapping bookmarks and aligned and supported on flat surface box. Then, with knee extended, subject flexes spine with head between arms up to the maximum range of motion, remaining static for about two seconds, while evaluator carry out reading on scale. Measures will be carried out three times, adopting highest value achieved. The cutoff points for flexibility will be proposed by project Sport Brazil (PROESP-BR), which classifies results into three categories: below (<23 cm), in (23-28 cm) and above (> 28 cm ) health and fitness area.
Flexibility parameters in hypertensive individuals | Baseline
  To describe flexibility parameters accordingly to Canadian Standardized Test of Fitnnes in hypertensive subjects.
Composite Outcome measure - association between AMBP parameters and Global Muscle Strength | Baseline
  Verify whether there is an association between blood pressure parameters and Global Muscle Strength changings
Composite Outcome measure - association between AMBP parameters and Respiratory Muscle Strength | Baseline
  Verify whether there is an association between blood pressure parameters and Respiratory Muscle Strength changings
Composite Outcome measure - association between AMBP parameters and functional capacity | Baseline
  Verify whether there is an association between blood pressure parameters and functional capacity changings
Composite Outcome measure - association between double product parameters and Global Muscle Strength | Baseline
  Verify whether there is an association between double product parameters and Global Muscle Strength changings
Composite Outcome measure - association between double product parameters and Respiratory Muscle Strength | Baseline
  Verify whether there is an association between double product parameters and Respiratory Muscle Strength changings
Composite Outcome measure - association between double product parameters and functional capacity | Baseline
  Verify whether there is an association between double product parameters and functional capacity changings

CONTACTS AND LOCATIONS:
Overall Officials: ANA MARICE T LADEIA, Doctorade, Principal Investigator — ESCOLA BAHIANA DE MEDICINA E SAÚDE PÚBLICA
Locations (1):
- Escola Bahiana de Medicina E Saúde Pública, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kavounoudias A, Roll R, Roll JP. The plantar sole is a 'dynamometric map' for human balance control. Neuroreport. 1998 Oct 5;9(14):3247-52. doi: 10.1097/00001756-199810050-00021. PMID 9831459
- [Background] Ribot-Ciscar E, Roll JP. Ago-antagonist muscle spindle inputs contribute together to joint movement coding in man. Brain Res. 1998 Apr 27;791(1-2):167-76. doi: 10.1016/s0006-8993(98)00092-4. PMID 9593876
- [Background] Villechevrolle, O. Influence des semelles of reprogrammation posturale globale sur les tests oculomoteurs réalisés sur une des sujets présentant disfonction cranio-mandibulaire.Thèse, Nantes, 1994a
- [Background] Villechevrolle, O. Influence des semelles of reprogrammation posturale globale sur le test de Fukuda. Diplôme d'Université mémoire of the Parodontologie et d'occluso, Nantes, 1994b.
- [Background] Mallong SP. Étude prospective longitudinal suivi par of pacientes douloureux au cours d'une Reprogrammation posturale Globale (RPG). Résonances Européennes du Rachis. 2006; 14 (42): 1753-6.
- [Background] Brazilian Society of Cardiology / Brazilian Society of Hypertension / Brazilian Society of Nephrology. VI Brazilian Guidelines on Hypertension. Arq Bras Cardiol 2010; 95 (1 suppl.1): 1-51
- [Background] Ferreira SR, Moura EC, Malta DC, Sarno F. Frequency of arterial hypertension and associated factors: Brazil, 2006. Rev Saude Publica. 2009 Nov;43 Suppl 2:98-106. doi: 10.1590/s0034-89102009000900013. English, Portuguese. PMID 19936504
- [Background] Piccini RX, Facchini LA, Tomasi E, Siqueira FV, Silveira DS, Thume E, Silva SM, Dilelio AS. Promotion, prevention and arterial hypertension care in Brazil. Rev Saude Publica. 2012 Jun;46(3):543-50. doi: 10.1590/s0034-89102012005000027. Epub 2012 Apr 17. English, Portuguese. PMID 22510974
- [Background] Lopes MC, Marcon SS. [Arterial hypertension in the family: the need for family care]. Rev Esc Enferm USP. 2009 Jun;43(2):343-50. doi: 10.1590/s0080-62342009000200013. Portuguese. PMID 19655675
- [Background] Schulz RB, Rossignoli P, Correr CJ, Fernandez-Llimos F, Toni PM. Validation of the short form of the Spanish hypertension quality of life questionnaire (MINICHAL) for Portuguese (Brazil). Arq Bras Cardiol. 2008 Feb;90(2):127-31. doi: 10.1590/s0066-782x2008000200010. English, Portuguese. PMID 18392385
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Colne P, Frelut ML, Peres G, Thoumie P. Postural control in obese adolescents assessed by limits of stability and gait initiation. Gait Posture. 2008 Jul;28(1):164-9. doi: 10.1016/j.gaitpost.2007.11.006. Epub 2008 Jan 10. PMID 18191568
- [Result] Roll JP, Bergenheim M, Ribot-Ciscar E. Proprioception Muscle afferents Sensory coding
- [Result] Kavounoudias A, Roll R, Roll JP. Foot sole and ankle muscle inputs contribute jointly to human erect posture regulation. J Physiol. 2001 May 1;532(Pt 3):869-78. doi: 10.1111/j.1469-7793.2001.0869e.x. PMID 11313452
- [Result] Roll R, Kavounoudias A, Roll JP. Cutaneous afferents from human plantar sole contribute to body posture awareness. Neuroreport. 2002 Oct 28;13(15):1957-61. doi: 10.1097/00001756-200210280-00025. PMID 12395099
- [Result] Grassi G, Seravalle G, Quarti-Trevano F. The 'neuroadrenergic hypothesis' in hypertension: current evidence. Exp Physiol. 2010 May;95(5):581-6. doi: 10.1113/expphysiol.2009.047381. Epub 2009 Dec 11. PMID 20008032
- [Result] Fisher JP, Fadel PJ. Therapeutic strategies for targeting excessive central sympathetic activation in human hypertension. Exp Physiol. 2010 May;95(5):572-80. doi: 10.1113/expphysiol.2009.047332. Epub 2010 Mar 19. PMID 20304932
- [Result] Tsioufis C, Kordalis A, Flessas D, Anastasopoulos I, Tsiachris D, Papademetriou V, Stefanadis C. Pathophysiology of resistant hypertension: the role of sympathetic nervous system. Int J Hypertens. 2011 Jan 20;2011:642416. doi: 10.4061/2011/642416. PMID 21331155
- [Result] Bruno RM, Ghiadoni L, Seravalle G, Dell'oro R, Taddei S, Grassi G. Sympathetic regulation of vascular function in health and disease. Front Physiol. 2012 Jul 24;3:284. doi: 10.3389/fphys.2012.00284. eCollection 2012. PMID 22934037
- [Result] Cavalcante MA, Bombig MT, Luna Filho B, Carvalho AC, Paola AA, Povoa R. Quality of life of hypertensive patients treated at an outpatient clinic. Arq Bras Cardiol. 2007 Oct;89(4):245-50. doi: 10.1590/s0066-782x2007001600006. English, Portuguese. PMID 17992381
- See also: List of validated instruments of BP assessment — http://www.dableducational.org/sphygmomanometers/devices_2_sbpm.html